CLINICAL TRIAL: NCT00923637
Title: Feasibility of Administering Adjuvant Chemotherapy of Pemetrexed Followed by Pemetrexed/Oxaliplatin Immediately Post-VATS in Patients With Completely Resected NSCLC
Brief Title: Pemetrexed Plus Oxaliplatin as Adjuvant Chemotherapy for Radically Resected Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Jianxing He, MD, FACS, The First Affiliated Hospital of Guangzhou Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20090601A
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; video assisted thoracic surgery; Adjuvant chemotherapy; Pemetrexed; Oxaliplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pemetrexed/Oxaliplatin — In the first cycle, patients received Pemetrexed 500 mg/m2 (i.v. infusion over 10 minutes) on day 1 of a 21-day cycle. From 2nd cycle, patients received pemetrexed 500 mg/m2 (i.v. infusion over 10 minutes) then oxaliplatin 120 mg/m2 (i.v. infusion over 120 minutes) on day 1 of a 21-day cycle. Study drug administration is to begin on d14 to d28 after R0 resection of the tumor. A total of three cycles is intended for patients with stage IB NSCLC, and four cycles for II-IIIA NSCLC, respectively.
  Other Names: Pemtrexed (Alimta); Oxaliplatin (Eloxatin)

SUMMARY:
The main purpose of this phase II trial is to evaluate the clinical feasibility-in terms of patients without dose limiting toxicities or premature treatment withdrawal or death-of administering adjuvant chemotherapy of pemetrexed followed by pemetrexed/oxaliplatin immediately post-video-assisted thoracic surgery (VATS) in patients with completely resected Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for the largest number of cancer deaths annually, worldwide. (Ferlay et al, 2007) Of these, about 30% are early stage patients (stage I and II). For this group of patients, radical surgery with mediastinal lymph node dissection has been the mainstay of therapy with a reasonable curative option. However, 5-year survival rates for patients with pathologically staged IA-IIB disease are ranging from 67% to 39%. (Mountain et al, 1997) Following surgery, distant recurrence is the most common form of relapse and eventual cause of death. Assuming that these recurrences are due to occult micrometastases at the time of surgery, trials on adjuvant systemic therapy have been performed in an attempt to reduce the risk of recurrence and to improve survival.

In some of the recently published trials a clear benefit of adjuvant chemotherapy in early stage NSCLC could not be achieved. (Tada et al, 2004; Scagliott et al, 2003; Waller et al, 2004) In marked contrast to these studies, three recent, big randomized trials on early stage NSCLC patients with modern platin-based two-drug chemotherapy-regimens revealed a significant advantage for overall or relapse free survival for chemotherapeutically treated patients. (Arriagada et al, 2004; Winton et al, 2005; Douillard et al, 2006) The majority of patients in the adjuvant treatment setting received a combination of cisplatin and vinorelbine. A pooled analysis of five big randomized studies demonstrated that adjuvant cisplatin-based chemotherapy significantly improves survival in patients with NSCLC (overall HR of death 0.89, P=0.005) corresponding to a 5-year absolute benefit of 5.4% from chemotherapy. (Pignon et al, 2008) However, toxicity and inadequate dose delivery have been critical issues in all trials performed so far. Grade 3/4 toxicities are observed up to 73% with rates of neutropenic fever up to 7%. Up to 77% of the patients had at least one dose reduction or omission and 55% required one dose delay or more, most related to neutropenia. (Pisters et al, 2005; Winton et al, 2005)

There are few data in the literature about how soon after surgery a patient begins adjuvant chemotherapy, although most trials seem to start after a post-surgical interval of 4-6 weeks. A recent study reported that 26 patients, who underwent thoracoscopic (video-assisted thoracic surgery, VATS) lobectomy, receiving chemotherapy, 73% completed a full course on schedule and 85% received all intended cycles. (Nicastri et al, 2008) In another study, complete resection was performed by thoracotomy in 43 patients and by thoracoscopy in 57 patients, compared with thoracotomy, patients undergoing thoracoscopic lobectomy had significantly fewer delayed (18% versus 58%, P < 0.001) and reduced (26% versus 49%, P = 0.02) chemotherapy doses. A higher percentage of patients undergoing thoracoscopic resection received 75% or more of their planned adjuvant regimen without delayed or reduced doses (61% versus 40%, P = 0.03). There were no significant differences in time to initiation of chemotherapy or toxicity. (Peterson et al, 2007) In comparison, the Cancer and Leukemia Group B trial 9633 reported that 57% of patients received full-dose chemotherapy (Strauss et al, 2008) and the Intergroup JBR.10 trial reported that 55% of patients had at least 1 dose delay. (Winton et al, 2005) Approximately 34% of patients in the Adjuvant Lung Project Italy series chemotherapy wing received all scheduled doses without adjustment or delay; 69% completed their treatments with or without adjustments or delay.(Scagliotti et al, 2003) It is conceivable that patients who undergo VATS may have a quicker recovery and in general more strength to tolerate chemotherapy. There are theoretic survival benefits to starting chemotherapy immediately after surgery because the body's tumor burden should be lowest, and tumor growth fastest, at this time. Thus, chemotherapy administered immediately post-surgery would be most effective, assuming that wound healing is adequate. (Nicastri et al, 2008)

Pemetrexed, a multi-target folate antimetabolite, shows clear activity in non-small cell lung cancer. In a phase III study for patients with previously treated advanced non-small cell lung cancer, the efficacy of single-agent pemetrexed, as determined by overall survival, was similar to that of docetaxel. (Hanna et al, 2004) The combination of oxaliplatin and pemetrexed has been of particular interest because it has demonstrated both good efficacy and a tolerable side effect profile. Oxaliplatin is a diaminocyclohexane-containing platinum compound that inhibits DNA replication and transcription by forming DNA adducts. Its mechanism of action is similar to that of the classic platinum drugs, but molecular pharmacology studies suggest that oxaliplatin represents a distinct family of platinum compounds. It has a different cytotoxicity profile from cisplatin and can be safely given in the outpatient setting without hydration therapy. (Raymond et al, 1998) Moreover, oxaliplatin appears to interact synergistically with pemetrexed. (Raymond et al, 2002) Phase I studies evaluated pemetrexed plus oxaliplatin in patients with solid tumors, and showed the regimen was efficacious and well tolerated. (Misset et al, 2004) The combination of oxaliplatin and pemetrexed was compared with carboplatin and pemetrexed as first-line therapy for advanced NSCLC in a randomized phase II study. Response rates were 27 and 33%, respectively, and not statistically different. However, toxicity in the oxaliplatin/pemetrexed arm was quite low, this doublet can be delivered easily and is well tolerated. Furthermore, it results in a 7.3% rate of grade 3/4 neutropenia only and the incidence of febrile neutropenia was 2.4%. Dose reductions occur only in 2.6% cycles. Patients received 95.3% and 100% of the planned weekly mean doses of pemetrexed and oxaliplatin, respectively. (Scagliotti et al, 2005)

Therefore, it seems reasonable to test a less toxic regimen also in early stages after complete (R0) resection of the tumor, where reduced toxicities might improve the feasibility of drug delivery, compliance and the convenience of treatment for the patient and hence perhaps improve survival. The main purpose of this phase II trial is to evaluate the clinical feasibility-in terms of patients without dose limiting toxicities or premature treatment withdrawal or death-of administering adjuvant chemotherapy of pemetrexed followed by pemetrexed/oxaliplatin immediately post-VATS in patients with completely resected NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with completely resected stage IB (> 4 cm), II, or IIIA non-squamous NSCLC by VATS. Patient must be enrolled and begin therapy within 4 weeks from the date of complete surgical resection.
* Fresh tissue must be available for genomics expression profiling.
* ECOG performance status of 0 or 1.
* No prior chemotherapy, radiation therapy, or biologic/targeted therapy within the last 5 years. Prior therapy with low dose methotrexate or similar medications is allowed if therapy used to treat non-malignant conditions.
* Age ≥ 18 years.
* No previous or concomitant malignancy in the past 5 years other than curatively-treated carcinoma in situ of the cervix, or basal cell or squamous cell carcinoma of the skin.
* No other serious medical or psychiatric illness.
* Signed informed consent.
* Required laboratory data within one week of enrollment:

  * ANC or AGC ≥ 1500 per uL;
  * Platelets ≥ 100,000 per uL;
  * Total bilirubin ≤ 1.5 mg/dL;
  * Creatinine < 2 mg/dL, creatinine clearance ≥ 45 mL/min;
  * SGOT/SGPT ≤ 1.5× ULN.
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 7 days prior to or at the time of enrollment based on a serum pregnancy test.
* Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determined by the patient and their health care team, during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent administration of any other anti-tumor therapy.
* Inability to comply with protocol or study procedures.
* Active infection requiring IV antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant systemic disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications.
* Contraindication to corticosteroids.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Unwillingness to stop taking herbal supplements while on study.
* Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study entry and throughout study enrollment as the distribution of pemetrexed in this fluid space is not fully understood.
* Inability to discontinue administration of aspirin at a dose > 1300 mg/day or other long acting, non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam). Moderate dose ibuprofen may be continued.
* Female patients that are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
To determine the clinical feasibility rate (CFR) of 4 cycles of adjuvant chemotherapy with pemetrexed followed by pemetrexed/oxaliplatin in patients with NSCLC stage IB, IIA, IIB and IIIA after a postsurgical interval of 2-4 weeks. | Every 21 days

SECONDARY OUTCOMES:
To determine the time to treatment failure, the relapse free survival, the overall survival, the distant metastases free survival, local relapse free survival, the localization of relapse. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Li SB, He JX, Chen HZ, Ge LH, Wei B, Yin WQ, Cheng XY, Liu J, Xu X. [Injection of activated carbon nanoparticles for guiding lymphadenectomy during minimal invasive surgery in lung cancer]. Zhonghua Zhong Liu Za Zhi. 2008 Mar;30(3):228-30. Chinese. PMID 18756943